CLINICAL TRIAL: NCT00081029
Title: A Multicentre Randomised Study Of Parotid Sparing Intensity Modulated Radiotherapy Versus Conventional Radiotherapy In Patients With Head And Neck Cancer
Brief Title: Parotid-Sparing Intensity-Modulated Radiation Therapy Compared With Conventional Radiation Therapy in Treating Patients With Oropharyngeal or Hypopharyngeal Cancer Who Are at High Risk of Radiation-Induced Xerostomia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000358803; ICR-PARSPORT; EU-20304; ISRCTN48243537; MREC-03679
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2008-03

CONDITIONS: Head and Neck Cancer; Radiation Toxicity; Xerostomia
Keywords: xerostomia; radiation toxicity; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Xerostomia; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

INTERVENTIONS:
Procedure: management of therapy complications
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Intensity-modulated radiation therapy delivers thin beams of radiation of different strengths directly to the tumor from many angles. This type of radiation therapy may reduce damage to the parotid (salivary) glands, prevent xerostomia (dry mouth), and improve quality of life. It is not yet known whether intensity-modulated radiation therapy is more effective than conventional radiation therapy in preventing xerostomia and improving quality of life in patients who have throat cancer.

PURPOSE: This randomized phase III trial is studying intensity-modulated radiation therapy to see how well it works compared to conventional radiation therapy in treating patients with oropharyngeal or hypopharyngeal cancer who are at risk of developing xerostomia caused by radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the proportion of patients with oropharyngeal or hypopharyngeal cancer with xerostomia of ≥ grade 2 at one year after treatment with parotid-sparing intensity-modulated radiotherapy vs conventional radiotherapy.

Secondary

* Compare the degree of xerostomia by quantitative measurements of stimulated and unstimulated salivary flow in patients treated with these regimens.
* Compare quality of life in patients treated with these regimens.
* Compare local and regional tumor control, time to tumor progression, and overall survival of patients treated with these regimens.
* Compare acute and late side effects of these regimens in these patients.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to participating center and site of disease (oropharynx vs hypopharynx). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo parotid-sparing intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks.
* Arm II: Patients undergo conventional radiotherapy once daily, 5 days a week, for 6 weeks.

Salivary flow measurements are performed at baseline, at week 4 during radiotherapy, and then at 2 weeks and at 3, 6, 12, and 24 months after the completion of radiotherapy.

Quality of life is assessed at baseline, at 2 weeks, and then at 3, 6, 12, 18, and 24 months after the completion of radiotherapy.

Patients are followed monthly for 1 year, every 2 months for 1 year, and then every 6 months for 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 84 patients (42 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed oropharyngeal or hypopharyngeal cancer

  * Squamous cell or undifferentiated carcinoma
  * Stage T1-4, N0-3, M0 disease
* Primary tumor requiring radical radiotherapy with parallel opposed lateral fields and bilateral cervical lymph node irradiation

  * Radiotherapy is either the primary therapy or post-operative (adjuvant irradiation) treatment
* High-risk for radiation-induced xerostomia with conventional radiotherapy due to irradiation of the majority of both parotid glands* NOTE: *Estimated mean dose to both parotid glands is greater than 24 Gy by conventional radiotherapy
* No bilateral N3 nodal disease
* No huge primary tumor (exceeding 10 cm in diameter)
* No contralateral lymphadenopathy adjacent to or involving contralateral parotid gland making parotid sparing impossible
* No tumor at the base of the tongue where sparing of contralateral parapharyngeal space is contraindicated

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to undergo quality of life and salivary flow measurements (dependent on cognitive aptitude and long availability)
* Able to complete self-assessed quality of life questionnaire
* No prior or concurrent illness that would preclude study participation
* No pre-existing salivary gland pathology interfering with saliva production
* No other prior malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior neoadjuvant chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to the head and neck region
* No concurrent brachytherapy

Surgery

* See Disease Characteristics

Other

* No concurrent prophylactic amifostine or pilocarpine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2004-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients suffering xerostomia ≥ grade 2 by LENT/SOMA late toxicity scale at 1 year

SECONDARY OUTCOMES:
Degree of xerostomia by salivary flow at 1 year
Xerosomia-related quality of life by Modified Xerostomia questionnaire at 1 year
Quality of Life by EORTC QLQ C30 v.3.0 and QLQ-H&N35 questionnaires at 1 year
Local and regional tumor control by a quantitative description of sites of relapse at 1 year
Time to tumor progression at 1 year
Overall survival at 1 year
Acuteside effects of radiotherapy by NCI CTCAE scale v. 3.0 at 1 year
Late side effects of radiotherapy by NCI CTCAE scale v3.0, LENT SOMA and RTOG at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nutting, Study Chair — Royal Marsden NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - Addenbrooke's Hospital, Cambridge, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Barts and the London School of Medicine, London, England
  - Royal Marsden - London, London, England
  - University College Hospital - London, London, England
  - Christie Hospital, Manchester, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England

REFERENCES:
- [Result] Nutting CM, Morden JP, Harrington KJ, Urbano TG, Bhide SA, Clark C, Miles EA, Miah AB, Newbold K, Tanay M, Adab F, Jefferies SJ, Scrase C, Yap BK, A'Hern RP, Sydenham MA, Emson M, Hall E; PARSPORT trial management group. Parotid-sparing intensity modulated versus conventional radiotherapy in head and neck cancer (PARSPORT): a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2011 Feb;12(2):127-36. doi: 10.1016/S1470-2045(10)70290-4. Epub 2011 Jan 12. PMID 21236730
- [Result] Clark CH, Hansen VN, Chantler H, Edwards C, James HV, Webster G, Miles EA, Guerrero Urbano MT, Bhide SA, Bidmead AM, Nutting CM; PARSPORT Trial Management Group. Dosimetry audit for a multi-centre IMRT head and neck trial. Radiother Oncol. 2009 Oct;93(1):102-8. doi: 10.1016/j.radonc.2009.04.025. PMID 19596158
- [Result] Clark CH, Miles EA, Urbano MT, Bhide SA, Bidmead AM, Harrington KJ, Nutting CM; UK PARSPORT Trial Management Group collaborators. Pre-trial quality assurance processes for an intensity-modulated radiation therapy (IMRT) trial: PARSPORT, a UK multicentre Phase III trial comparing conventional radiotherapy and parotid-sparing IMRT for locally advanced head and neck cancer. Br J Radiol. 2009 Jul;82(979):585-94. doi: 10.1259/bjr/31966505. Epub 2009 Mar 30. PMID 19332518